CLINICAL TRIAL: NCT00700050
Title: Modulation by Sex Hormones of Inflammation and Susceptibility to Pseudomonas Aeruginosa in Cystic Fibrosis Airways - A Pilot Study
Brief Title: Modulation by Sex Hormones of Inflammation and Susceptibility to Pseudomonas Aeruginosa in Cystic Fibrosis Airways
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Neil Sweezey, Staff Respirologist, The Hospital for Sick Children
Other Study IDs: 1000011620
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Sex hormones; Pseudomonas aeruginosa; Paediatrics
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Saline Solution, Hypertonic; Sodium Chloride; Inhalation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CF Females: CF females, 14 - 28 years old, sexually mature, with regular menstrual cycles, not on contraceptive Pill. No intervention is being tested - subjects studied with normal menstrual variations in serum hormone levels. Hypertonic saline may be used to induce sputum production by subjects who are otherwise unable to produce a satisfactory sputum sample.
  Interventions: Drug: Hypertonic saline
- Non-CF Females: Non-CF control females, 14 - 28 years old, sexually mature, with regular menstrual cycles, not on contraceptive Pill. No intervention is being tested - subjects studied with normal menstrual variations in serum hormone levels. Hypertonic saline may be used to induce sputum production by subjects who are otherwise unable to produce a satisfactory sputum sample.
  Interventions: Drug: Hypertonic saline
- CF Males: CF males, 14 - 28 years old. No intervention is being tested. Hypertonic saline may be used to induce sputum production by subjects who are otherwise unable to produce a satisfactory sputum sample.
  Interventions: Drug: Hypertonic saline
- Non-CF males: Non-CF control males, 14 - 28 years old. No intervention is being tested. Hypertonic saline may be used to induce sputum production by subjects who are otherwise unable to produce a satisfactory sputum sample.
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Hypertonic saline — Subjects will be asked to expectorate sputum samples. If necessary to achieve this, subjects will inhale wet-nebulized 3% saline for up to 7 minutes each for up to 3 cycles.
  Other Names: Sodium chloride, inhalation;
  Groups: CF Females
Drug: Hypertonic saline — Subjects will be asked to expectorate sputum samples. If necessary to achieve this, subjects will inhale wet-nebulized 3% saline for up to 7 minutes each for up to 3 cycles.
  Other Names: Sodium chloride, inhalation
  Groups: Non-CF Females
Drug: Hypertonic saline — Subjects will be asked to expectorate sputum samples. If necessary to achieve this, subjects will inhale wet-nebulized 3% saline for up to 7 minutes each for up to 3 cycles.
  Other Names: Sodium chloride, inhalation
  Groups: CF Males
Drug: Hypertonic saline — Subjects will be asked to expectorate sputum samples. If necessary to achieve this, subjects will inhale wet-nebulized 3% saline for up to 7 minutes each for up to 3 cycles.
  Other Names: Sodium chloride, inhalation
  Groups: Non-CF males

SUMMARY:
The general objective is to elucidate the mechanisms whereby sex hormones may modulate the severity of respiratory disease. An important component of this proposal is a systematic and intensive approach to characterize how the cellular and cytokine components of airway inflammation respond to fluctuations in sex hormone levels.

The effects of menstrual fluctuations in levels of sex hormones on inflammation and bacterial load in respiratory secretions of CF patients will also be determined.

DETAILED DESCRIPTION:
Most CF patients die because of chronic lung infection with P. aeruginosa, chronic inflammation and progressive airway damage. Agents that reduce inflammation or enhance airway antibacterial defences hold potential therapeutic value. Therefore, there is considerable current interest in identifying and stimulating the activities of these agents. Although sex hormones are generally acknowledged to modulate respiratory inflammation, the downstream mechanism of such action remains incompletely understood.

We have identified three antimicrobial peptides (AMPs), responsive to sex hormone in the CF human respiratory tract, including one (LTF) with known activity against P. aeruginosa biofilm formation. Our preliminary results show additive activity of LTF and STH against P. aeruginosa biofilm formation, and that LTF and STH also inhibit attachment of P. aeruginosa to airway epithelial cells. Taken together, these findings are consistent with the concept that female sex hormones exert their negative effect on the CF lung, in part, by reducing the levels of these AMPs in the airway. The next step is to determine if female sex hormones alter airway inflammation and infection or AMP levels in the respiratory secretions of CF patients.

ELIGIBILITY:
Inclusion Criteria:

FEMALES WITH CF

* Sexually mature female CF patients followed at the Toronto CF Clinics of The Hospital for Sick Children (adolescents) or St. Michael's Hospital (adults)
* 14-28 years of age
* Diagnosis of CF is based on a typical clinical picture and confirmed by repeated sweat chloride values > 60 mEq/L as determined by pilocarpine ionophoresis (minimum 100mg sweat)
* Have regular, normal menses
* Able to give consent on her own behalf

FEMALES WITHOUT CF

* Sexually mature females
* 14-28 years of age
* Have regular, normal menses
* Able to give consent on her own behalf

MALES WITH CF

* Sexually mature male CF patients followed at the Toronto CF Clinics of The Hospital for Sick Children (adolescents) or St. Michael's Hospital (adults)
* 14-28 years of age
* Diagnosis of CF is based on a typical clinical picture and confirmed by repeated sweat chloride values > 60 mEq/L as determined by pilocarpine ionophoresis (minimum 100mg sweat)
* Able to give consent on his own behalf

MALES WITHOUT CF

* Sexually mature males
* 14-28 years of age
* Able to give consent on his own behalf

Exclusion Criteria:

* Is a smoker
* Has had an upper respiratory tract infection within the preceding two weeks
* Is taking systemic oral contraceptive therapy
* Is pregnant
* Has used furosemide or amiloride or had a pulmonary exacerbation in the previous month (Acute exacerbations are defined as 3 or more of the following symptoms or signs: increased cough, change in volume, colour or thickness of the sputum, fever, hemoptysis, increased shortness of breath, change in their chest radiograph or a fall in pulmonary function (FEV1) of >10% from baseline)
* Unable to give consent on his/her own behalf

Ages: 14 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The primary study population are sexually mature cystic fibrosis (CF) females with regular natural menstrual cycles. For some measurements, they serve as their own controls. For other measurements, there are up to three control groups: non-CF females, CF males and non-CF males.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2014-07-29 (Actual); Study Completion 2014-07-29 (Actual)

PRIMARY OUTCOMES:
Presence of inflammatory markers (cytokines, white blood cells), levels of LTF, STH and PIP. Serum levels of estrogen (E), progesterone (P), luteinizing hormone (LH) and follicle stimulating hormone (FSH) will be determined in female human subjects | For the female patients the visits will be timed so that one measure is taken in the luteal phase of their menstrual cycle and the other is taken during the follicular phase. Male patients will be asked to come to measure these levels two weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sweezey, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada